CLINICAL TRIAL: NCT03607305
Title: Impact of Biliopancreatic Limb Lenght on Long-term Weight Loss After Roux-en-Y Gastric
Brief Title: Impact of Biliopancreatic Limb Lenght on Long-term Weight Loss After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGUE 2012-12
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP limb 70cm (Active Comparator): Patients underwent a RYGB with a biliopancreatic limb of 70cm
  Interventions: Procedure: BP limb 70cm
- BP limb 120cm (Experimental): Patients underwent a RYGB with a biliopancreatic limb of 120cm
  Interventions: Procedure: BP limb 120cm

INTERVENTIONS:
Procedure: BP limb 70cm — Performance of RYGB with a BP limb of 70cm
  Arms: BP limb 70cm
Procedure: BP limb 120cm — Performance of RYGB with a BP limb of 120cm
  Arms: BP limb 120cm

SUMMARY:
Patients were randomly assigned into 2 groups: those patients undergoing RYGB with a BPL of 70cm and those ones undergoing RYGB with a BPL of 120 cm.

Excess BMI loss 5 years after surgery was investigated

DETAILED DESCRIPTION:
Patients were randomly assigned into 2 groups: those patients undergoing Roux-en-Y gastric bypass with a biliopancreatic limb of 70cm and those ones undergoing Roux-en-Y gastric bypass with a biliopancreatic limb of 120 cm. Alimentary limb was constant in both groups (150cm).

Excess BMI loss 5 years after surgery was investigated

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity
* Age older than 18 years

Exclusion Criteria:

* Patients undergoing other bariatric techniques than RYGB
* Patients undergoing RYGB with different BPL or AL lengths than that reported for this study
* Any other surgical procedure added to the bariatric surgery
* Impossibility to comply with pre-established clinical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 5 years after surgery
  Weight loss was evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, Principal Investigator — HOSPITAL REY JUAN CARLOS

REFERENCES:
- [Derived] Ruiz-Tovar J, Vorwald P, Gonzalez-Ramirez G, Posada M, Salcedo G, Llavero C, Garcia-Olmo D. Impact of Biliopancreatic Limb Length (70 cm vs 120 cm), with Constant 150 cm Alimentary Limb, on Long-Term Weight Loss, Remission of Comorbidities and Supplementation Needs After Roux-En-Y Gastric Bypass: a Prospective Randomized Clinical Trial. Obes Surg. 2019 Aug;29(8):2367-2372. doi: 10.1007/s11695-019-03717-7. PMID 31104282